CLINICAL TRIAL: NCT04768296
Title: A Phase II, Open-label, Single-arm Study of Berzosertib (M6620) in Combination With Topotecan in Participants With Relapsed Platinum-resistant Small-Cell Lung Cancer (DDRiver SCLC 250)
Brief Title: Berzosertib + Topotecan in Relapsed Platinum-Resistant Small-Cell Lung Cancer (DDRiver SCLC 250)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: EMD Serono Research & Development Institute, Inc. (Industry)
Collaborators: Merck KGaA, Darmstadt, Germany (Industry)
Responsible Party: Sponsor
Organization: EMD Serono (Industry)
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: MS201923_0050; 2020-004231-25 (EudraCT Number)
Record Dates: First submitted 2021-02-19; First posted 2021-02-24 (Actual); Results first posted 2024-09-26 (Actual); Last update posted 2024-09-26 (Actual); Status verified 2024-08

CONDITIONS: Small-cell Lung Cancer
Keywords: M6620; Berzosertib; Solid Tumor; Topotecan; Ataxia telangiectasia mutated and Rad3-related; Platinum-resistant Small-Cell Lung Cancer; DDRiver
MeSH Terms: conditions — Small Cell Lung Carcinoma; Hereditary Sensory and Autonomic Neuropathies | interventions — berzosertib; Topotecan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Safety run-in Part (Dose Level1 [DL 1]): Berzosertib 105 mg/m^2 + Topotecan 1.25 mg/m^2 (Experimental): Participants received Berzosertib at a dose of 105 milligrams per square meter (mg/m^2 ) intravenously on Day 2 and Day 5 of each 21-daycycle in combination with Topotecan at a dose of 1.25mg/m^2 intravenously on Days1 through 5 of each 21-day cycle in DL1 of safety run-in part until disease progression or other criteria for study intervention discontinuation are met.
  Interventions: Drug: Berzosertib; Drug: Topotecan
- Safety run-in Part (DL2) +Main Part: Berzosertib 210 mg/m^2 + Topotecan 1.25 mg/m^2 (Experimental): Participants received Berzosertib at a dose of 210 mg/m^2 intravenously on Day 2 and Day 5 of each 21-day cycle in combination with Topotecan at a dose of 1.25 mg/m^2 intravenously on Days 1 through 5 of each 21-day cycle in DL 1 and DL 2 of safety run-in part and main part until disease progression or other criteria for study intervention discontinuation are met.
  Interventions: Drug: Berzosertib; Drug: Topotecan

INTERVENTIONS:
Drug: Berzosertib — Participants received Berzosertib at a dose of 105 milligrams per square meter (mg/m^2 ) intravenously on Day 2 and Day 5 of each 21-day cycle until disease progression or other criteria for study intervention discontinuation are met.
  Other Names: M6620
  Arms: Safety run-in Part (Dose Level1 [DL 1]): Berzosertib 105 mg/m^2 + Topotecan 1.25 mg/m^2
Drug: Berzosertib — Participants received Berzosertib at a dose of 210 mg/m^2 intravenously on Day 2 and Day 5 of each 21-day cycle in DL2 of safety run-in part and main part until disease progression or other criteria for study intervention discontinuation are met.
  Other Names: M6620
  Arms: Safety run-in Part (DL2) +Main Part: Berzosertib 210 mg/m^2 + Topotecan 1.25 mg/m^2
Drug: Topotecan — Participants received Topotecan at a dose of 1.25 mg/m^2 intravenously on Days 1 through 5 of each 21-day cycle in DL1 and DL2 of safety run-in part and main part until disease progression or other criteria for study intervention discontinuation are met.

SUMMARY:
The main purpose of this study is to assess efficacy, safety, tolerability and pharmacokinetics (PK) of Berzosertib in combination with Topotecan in participants with relapsed, platinum-resistant small-cell lung cancer (SCLC). This study will be conducted in two parts: safety run-in part and main part. The safety run-in part will be conducted in Japan.

ELIGIBILITY:
Inclusion Criteria:

* Dose level 1 participants with histologically proven advanced solid tumors, for which no effective standard therapy exists, or standard therapy has failed or cannot be tolerated
* Dose level 1 participants with Eastern Cooperative Oncology Group Performance Status (ECOG PS) less than or equal to (<=) 1 and Karnofsky Scale greater than or equal to (>=) 70 percent (%)
* Dose level 2 and main part participants with ECOG PS <= 2 and Karnofsky Scale >= 60%
* Dose level 2 and main part participants with histologically confirmed SCLC
* Dose level 2 and main part participants with radiologically confirmed progression after first-line or chemoradiation platinum-based treatment (carboplatin or cisplatin), with or without immunotherapy, for treatment of limited or extensive stage SCLC, with a Platinum-free interval (PFI) less than (<) 90 days. The PFI is measured by the elapsed time from the last day of the regimen of a platinum-based treatment until the first day of documented disease progression
* Dose level 2 and main part participants with measurable disease according to Response Evaluation Criteria in Solid Tumors (RECIST) Version 1.1 (RECISTv1.1) at Screening. Evidence of measurable disease must be confirmed by the IRC prior to start of treatment
* Tumor tissue provision: archival (collected within 12 months before date of informed consent form [ICF]) signature for Screening) or fresh biopsy specimen, if medically feasible
* Have adequate hematologic and renal function
* Other protocol defined inclusion criteria could apply

Exclusion Criteria:

* Clinically relevant (that is [i.e.], active), uncontrolled intercurrent illness including, but not limited to, severe active infection including, severe acute respiratory syndrome coronavirus-2 infection/coronavirus disease 2019, immune deficiencies, uncontrolled diabetes, uncontrolled arterial hypertension, symptomatic congestive heart failure (New York Heart Association Classification greater than or equal to [>=] Class III), unstable angina pectoris, myocardial infarction, uncontrolled cardiac arrhythmia, cerebral vascular accident/stroke. Calculated corrected QT interval (QTc) average (using the Fridericia correction calculation) of greater than [>] 450 millisecond (msec) for males and > 470 msec for females. Any psychiatric illness/social situations that would limit compliance with study requirements
* Unstable brain metastases; however, participants with known brain metastases may be enrolled in this clinical study if they are clinically stable (without evidence of progression by imaging for at least 2 weeks prior to the first study intervention dose and any neurologic symptoms have returned to baseline), have no evidence of new brain metastases, and are on a stable or decreasing dose of steroids for at least 14 days prior to study intervention Participants with carcinomatous meningitis are excluded regardless of clinical stability. Screening central nervous system imaging is not mandatory
* Prior malignant disease within the last 3 years. Exceptions include fully resected basal cell carcinoma of the skin or squamous cell carcinoma of the skin, in situ cervical cancer, fully resected ductal carcinoma in situ of the breast, superficial or noninvasive bladder cancer, and Stage IA, Grade I endometrioid endometrial cancer with no myometrial invasion, that has undergone curative therapy. Participants with other localized malignancies treated with curative intent need to be discussed with the Medical Monitor
* Participants not recovered from adverse events (AEs) Grade > 1 from prior anticancer therapies, including surgeries. Exception: Grade 2 AEs not constituting a safety risk (for example [e.g.], alopecia), based on the Investigator's judgment; must consult with the medical Monitor prior to enrollment.
* Other protocol defined exclusion criteria could apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Actual)
Dates: Start 2021-03-29 (Actual); Primary Completion 2023-07-21 (Actual); Study Completion 2023-07-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Responsible, Study Director — Merck Healthcare KGaA, Darmstadt, Germany, an affiliate of Merck KGaA, Darmstadt, Germany
Locations (51):
- United States (12):
  - Providence Medical Foundation, Santa Rosa, California
  - St Joseph Heritage Healthcare, Santa Rosa, California
  - Cotton-O'Neil Clinical Research Center, Hematology and Oncology, Topeka, Kansas
  - National Cancer Institute, Bethesda, Maryland
  - Cancer & Hematology Centers of Western Michigan, Grand Rapids, Michigan
  - MidAmerica Cancer Care, Kansas City, Missouri
  - NJ Center for Cancer Research, Brick, New Jersey
  - Southeastern Medical Oncology Center, Goldsboro, North Carolina
  - FirstHealth of the Carolinas, Inc., Pinehurst, North Carolina
  - Summa Health, Akron, Ohio
  - Toledo Clinic, Toledo, Ohio
  - Millennium Physicians Association, LLP, Houston, Texas
- Belgium (5):
  - Centre Hospitalier de l'Ardenne, Arlon
  - Institut Jules Bordet - Department of Institut Jules Bordet, Brussels
  - Universitair Ziekenhuis Gent, Ghent
  - AZ Delta, Roeselare
  - CHU UCL Namur - Mont-Godinne, Yvoir
- China (9):
  - Beijing Cancer Hospital, Beijing
  - Jilin Cancer Hospital, Changchun
  - Sichuan Cancer Hospital, Chengdu
  - West China Hospital, Sichuan University, Chengdu
  - Jiangsu Province Hospital, Nanjing
  - Liaoning Cancer Hospital & Institute, Shenyang
  - Union Hospital of Tongji Medical College, Huazhong University of Science and Technology, Wuhan
  - The First Affiliated Hospital of Xi'an Jiaotong University, Xi'an
  - The First Affiliated Hospital of Zhejiang University school of medicine, Zhejiang
- France (6):
  - Institut Bergonié, Bordeaux
  - Centre Hospitalier Intercommunal de Créteil - Service de Pneumologie, Créteil
  - Hopital Albert Calmette - CHU Lille - service de pneumologie et immuno allergologie, Lille
  - CHU Poitiers - Hôpital la Milétrie - service d'oncologie médicale, Poitiers
  - CHU Nantes - Hôpital Guillaume et René Laënnec - Service de Pneumologie, Saint-Herblain
  - CHU de Strasbourg - Nouvel Hôpital Civil - Service de Pneumologie, Strasbourg
- Italy (5):
  - IRCCS Istituto Scientifico Romagnolo Per Lo Studio e La Cura Dei Tumori "Dino Amadori" - IRST, Meldola
  - Azienda Socio Sanitaria Territoriale Niguarda (Grande Ospedale Metropolitano Niguarda), Milan
  - Azienda Ospedaliero Universitaria Pisana (Presidio di Cisanello), Pisa
  - Istituto Nazionale Tumori Regina Elena IRCCS, Roma
  - Fondazione Policlinico Universitario Agostino Gemelli IRCCS - UOC Oncologia Medica, Rome
- Japan (7):
  - National Cancer Center Hospital, Chūōku
  - Kansai Medical University Hospital, Hirakata-shi
  - National Cancer Center Hospital East, Kashiwa-shi
  - Cancer Institute Hospital of JFCR, Kōtoku
  - Kindai University Hospital, Osaka
  - Kurume University Hospital, Osaka
  - Osaka Medical and Pharmaceutical University Hospital, Takatsuki-shi
- Spain (7):
  - Hospital Clinic de Barcelona, Barcelona
  - Hospital Universitari Vall d'Hebron, Barcelona
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Universitario La Paz, Madrid
  - Hospital Clinico Universitario Virgen de la Victoria - Oncology Service, Málaga
  - Hospital Universitario Virgen de la Victoria, Málaga
  - Hospital Universitario Virgen Macarena, Seville

IPD SHARING:
Plan to Share IPD: Yes
We are committed to enhancing public health through responsible sharing of clinical trial data. Following approval of a new product or a new indication for an approved product in both the US and European Union, the study sponsor and/or its affiliated companies will share study protocols, anonymized patient data and study level data, and redacted clinical study reports with qualified scientific and medical researchers, upon request, as necessary for conducting legitimate research. Further information on how to request data can be found on our website bit.ly/IPD21
Supporting Information: Study Protocol, SAP, CSR, Analytic Code
Time Frame: Within six months after the approval of a new product or a new indication for an approved product in both the United States and the European Union
Access Criteria: Qualified scientific and medical researchers can request the data. Such requests must be submitted in writing to the company's portal and will be internally reviewed regarding criteria for researchers' qualification and legitimacy of the research proposal.
URL: https://bit.ly/IPD21

REFERENCES:
- See also: Trial Awareness and Transparency website — https://clinicaltrials.emdgroup.com/en/trial-details/?id=MS201923_0050
- See also: US Medical Information website, Medical Resources — https://medical.emdserono.com/en_US/home.html
- See also: DDRiver website — http://www.DDRiver-trials.com

RESULTS

PARTICIPANT FLOW:
Groups:
- Safety run-in Part (Dose Level 1 [DL 1]): Berzosertib 105 mg/m^2 + Topotecan 1.25 mg/m^2: Participants received Berzosertib at a dose of 105 milligrams per square meter (mg/m^2 ) intravenously on Day 2 and Day 5 of each 21-day cycle in combination with Topotecan at a dose of 1.25 mg/m^2 intravenously on Days 1 through 5 of each 21-day cycle in DL1 of safety run-in part until disease progression or other criteria for study intervention discontinuation are met.
- Safety run-in Part (DL2) + Main Part: Berzosertib 210 mg/m^2 + Topotecan 1.25 mg/m^2: Participants received Berzosertib at a dose of 210 mg/m^2 intravenously on Day 2 and Day 5 of each 21-day cycle in combination with Topotecan at a dose of 1.25 mg/m^2 intravenously on Days 1 through 5 of each 21-day cycle in DL1 and DL2 of safety run-in part and main part until disease progression or other criteria for study intervention discontinuation are met.
Period: Overall Study
Arm/Group | Safety run-in Part (Dose Level 1 [DL 1]): Berzosertib 105 mg/m^2 + Topotecan 1.25 mg/m^2 | Safety run-in Part (DL2) + Main Part: Berzosertib 210 mg/m^2 + Topotecan 1.25 mg/m^2
Started | 3 | 73
Completed | 2 | 66
Not Completed | 1 | 7
Not completed — STOP LONG-TERM FOLLOW-UP AS PER SPONSOR'S DECISION | 1 | 7

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Safety run-in Part (Dose Level 1 [DL 1]): Berzosertib 105 mg/m^2 + Topotecan 1.25 mg/m^2 | Safety run-in Part (DL2) + Main Part: Berzosertib 210 mg/m^2 + Topotecan 1.25 mg/m^2 | Total
Number analyzed (Participants) | 3 | 73 | 76
Age, Continuous [Mean (Standard Deviation); unit: Years] | 51 (4) | 63 (7.8) | 62 (8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 16 | 17
  Male | 2 | 57 | 59
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 1
  Not Hispanic or Latino | 3 | 63 | 66
  Unknown or Not Reported | 0 | 9 | 9
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 3 | 19 | 22
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 1 | 1
  White | 0 | 42 | 42
  More than one race | 0 | 1 | 1
  Unknown or Not Reported | 0 | 10 | 10

OUTCOME MEASURES:

1. Primary Outcome: Main Part: Objective Response Rate According to Response Evaluation Criteria in Solid Tumors (RECIST) Version 1.1 as Assessed by Independent Review Committee (IRC)
Description: Objective response rate was defined as percentage of participants with either a confirmed complete response (CR) or partial response (PR) from first administration of study treatment to first observation of progressive disease (PD). CR: Disappearance of all target and non-target lesions. PR: At least a 30 percent (%) decrease in the sum of diameters of target lesions, taking as reference the baseline sum of their diameters, and no unequivocal progression of non-target lesions. PD: at least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on the study, or unequivocal progression of non-target lesions, or appearance of any new lesion.
Time Frame: Time from first administration of study treatment up to 27.7 months
Population: Full Analysis Set (FAS) included all participants who were administered at least 1 dose of berzosertib.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Safety run-in Part (DL2) + Main Part: Berzosertib 210 mg/m^2 + Topotecan 1.25 mg/m^2
Number analyzed (Participants) | 73
percentage of participants | 5.5 [1.5 to 13.4]

2. Primary Outcome: Safety Run-in Part: Number of Participants With Dose Limiting Toxicities (DLTs)
Description: DLT is defined as drug-related: Neutropenia Grade 4 for greater than (>) 7 days' duration; Febrile neutropenia (that is [i.e.] absolute neutrophil count less than (< ) 1000 per millimeter cube (mm^3) with single temperature of > 38.3°degree Celsius or a sustained temperature of greater than or equal to (>=) 38 degree Celsius for more than 1 hour; Infection (documented clinically or microbiologically) with Grades 3 or 4 neutropenia; Thrombocytopenia >= Grade 3; Grade >= 3 non-hematological AEs.
Time Frame: Up to Cycle 1 Day 21 (each cycle is of 21 days)
Population: DLT analysis set: all participants who were administered any dose of any study intervention in Safety Run-in Part in Japan and meet at least one of the following criteria: Received at least 80% of planned cumulative dose of study intervention during the DLT and completed the DLT period. The final decision on evaluability is made by the SMC; Experienced at least 1 DL T during the DLT period, regardless of the administered cumulative dose of study intervention and completion of the DLT period.
Measure: Count of Participants; unit: Participants
Groups:
- Safety run-in Part (DL 1): Berzosertib 105 mg/m^2 + Topotecan 1.25 mg/m^2: Participants received Berzosertib at a dose of 105 milligrams per square meter (mg/m^2 ) intravenously on Day 2 and Day 5 of each 21-day cycle in combination with Topotecan at a dose of 1.25 mg/m^2 intravenously on Days 1 through 5 of each 21-day cycle in safety run-in part until disease progression or other criteria for study intervention discontinuation are met.
Arm/Group | Safety run-in Part (DL 1): Berzosertib 105 mg/m^2 + Topotecan 1.25 mg/m^2 | Safety run-in Part (DL2) + Main Part: Berzosertib 210 mg/m^2 + Topotecan 1.25 mg/m^2
Number analyzed (Participants) | 3 | 3
Participants | 0 | 0

3. Primary Outcome: Safety Run-in Part: Number of Participants With Treatment-Emergent Adverse Events (TEAEs) and Treatment-Related TEAEs
Description: An adverse event (AE) is defined as any untoward medical occurrence in a participant or clinical study participant, temporally associated with the use of study intervention, whether considered related to the study intervention or not. A serious AE was an AE that resulted in any of the following outcomes: death; life threatening; persistent/significant disability/incapacity; initial or prolonged inpatient hospitalization; congenital anomaly/birth defect or was otherwise considered medically important. TEAEs were defined as events with onset date or worsening during the on-treatment period. TEAEs included both serious and non-serious TEAEs. Treatment-related TEAEs is defined as reasonably related to the study intervention.
Time Frame: Time from first administration of study treatment up to 27.7 months
Population: Safety (SAF) Analysis Set included all participants who were administered at least 1 dose of berzosertib.
Measure: Count of Participants; unit: Participants
Arm/Group | Safety run-in Part (DL 1): Berzosertib 105 mg/m^2 + Topotecan 1.25 mg/m^2 | Safety run-in Part (DL2) + Main Part: Berzosertib 210 mg/m^2 + Topotecan 1.25 mg/m^2
Number analyzed (Participants) | 3 | 3
Participants
  TEAEs | 3 | 3
  Treatment Related TEAEs | 3 | 3

4. Primary Outcome: Safety Run-in Part: Number of Participants With Clinically Significant Changes From Baseline in Vital Signs
Description: Vital signs included body temperature, heart rate, systolic and diastolic blood pressure and respiration rate. Number of participants with clinically significant changes from baseline in vital signs were reported. Clinical significance was decided by Investigator.
Time Frame: Time from first administration of study treatment up to 27.7 months
Population: Safety (SAF) Analysis Set included all participants who were administered at least 1 dose of berzosertib.
Measure: Count of Participants; unit: Participants
Arm/Group | Safety run-in Part (DL 1): Berzosertib 105 mg/m^2 + Topotecan 1.25 mg/m^2 | Safety run-in Part (DL2) + Main Part: Berzosertib 210 mg/m^2 + Topotecan 1.25 mg/m^2
Number analyzed (Participants) | 3 | 3
Participants | 0 | 0

5. Primary Outcome: Safety Run-in Part: Number of Participants With Clinically Significant Changes From Baseline in 12-Lead Electrocardiogram (ECG) Findings
Description: ECG parameters included PR interval, RR interval, QT interval, QRS duration, QTc intervals (derived using Fridericia's correction method) and heart rate. A 12-lead ECG was recorded with the participant in a supine position after a rest of at least 5 minutes using an ECG machine. Clinical significance was decided by investigator. Number of participants with clinically significant changes from baseline in 12-Lead ECGs were reported.
Time Frame: Time from first administration of study treatment up to 27.7 months
Population: Safety (SAF) Analysis Set included all participants who were administered at least 1 dose of berzosertib.
Measure: Count of Participants; unit: Participants
Arm/Group | Safety run-in Part (DL 1): Berzosertib 105 mg/m^2 + Topotecan 1.25 mg/m^2 | Safety run-in Part (DL2) + Main Part: Berzosertib 210 mg/m^2 + Topotecan 1.25 mg/m^2
Number analyzed (Participants) | 3 | 3
Participants | 0 | 0

6. Primary Outcome: Safety Run-in Part: Number of Participants With Clinically Significant Abnormalities in Laboratory Values Reported as Treatment Emergent Adverse Events (TEAEs)
Description: The laboratory measurements included hematology and biochemistry. Number of participants with clinically significant abnormalities with Grade greater than or equals to (>=) 3 in laboratory values reported as TEAEs as per National Cancer Institute Common Terminology Criteria for Adverse Events (NCI-CTCAE) v5.0 graded from Grade 1 to 5. Grade 1: Mild; Grade 2: Moderate; Grade 3: Severe; Grade 4: Life-threatening; Grade 5: Death. Clinically Significance was decided by investigator.
Time Frame: Time from first administration of study treatment up to 27.7 months
Population: Safety (SAF) Analysis Set included all participants who were administered at least 1 dose of berzosertib.
Measure: Count of Participants; unit: Participants
Arm/Group | Safety run-in Part (DL 1): Berzosertib 105 mg/m^2 + Topotecan 1.25 mg/m^2 | Safety run-in Part (DL2) + Main Part: Berzosertib 210 mg/m^2 + Topotecan 1.25 mg/m^2
Number analyzed (Participants) | 3 | 3
Participants
  Hematology | 0 | 3
  Biochemistry | 0 | 0

7. Secondary Outcome: Main Part: Duration of Response (DoR) According to Response Evaluation Criteria in Solid Tumors (RECIST) Version 1.1 as Assessed by Independent Review Committee (IRC)
Description: DoR was defined for participants with objective response, as the time from first documentation of objective response (Complete Response [CR] or Partial Response [PR]) to the date of first documentation of progression disease (PD) or death due to any cause, whichever occurred first. CR: Disappearance of all target and non-target lesions. PR: At least a 30 percent (%) decrease in the sum of diameters of target lesions, taking as reference the baseline sum of their diameters, and no unequivocal progression of non-target lesions. PD: at least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on the study, or unequivocal progression of non-target lesions, or appearance of any new lesion.
Time Frame: From first documented objective response to PD or death due to any cause, assessed up to 27.7 months
Population: FAS was used. Due to small number of participants with a response, data was not summarized; however, individual participant data is reported for this outcome measure. Here, "Overall Number of Participants Analyzed" = participants who were evaluable for this outcome measure and "number analyzed" = specific participants evaluated in the arm.
Measure: Number; unit: months
Arm/Group | Safety run-in Part (DL2) + Main Part: Berzosertib 210 mg/m^2 + Topotecan 1.25 mg/m^2
Number analyzed (Participants) | 4
months
  Participant 1: number analyzed (Participants) | 1
  Participant 1 | 8.5
  Participant 2: number analyzed (Participants) | 1
  Participant 2 | 2.8
  Participant 3: number analyzed (Participants) | 1
  Participant 3 | 2.6
  Participant 4: number analyzed (Participants) | 1
  Participant 4 | 2.1

8. Secondary Outcome: Main Part: Progression-free Survival (PFS) According to Response Evaluation Criteria in Solid Tumors (RECIST) Version 1.1 as Assessed by Independent Review Committee (IRC)
Description: PFS was defined as the time is defined as the time from first administration of study treatment to the date of the first documentation of PD or death due to any cause, whichever occurs first. PD: at least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on the study, or unequivocal progression of non-target lesions, or appearance of any new lesion.
Time Frame: Time from first administration of study treatment to the date of the first documentation of PD or death due to any cause, assessed up to 27.7 months
Population: Full Analysis Set (FAS) included all participants who were administered at least 1 dose of berzosertib.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Safety run-in Part (DL2) + Main Part: Berzosertib 210 mg/m^2 + Topotecan 1.25 mg/m^2
Number analyzed (Participants) | 73
months | 2.2 [1.5 to 2.7]

9. Secondary Outcome: Main Part: Overall Survival (OS)
Description: Overall survival is defined as the time from first administration of study treatment to the date of death.
Time Frame: Time from first administration of study treatment to the date of death, assessed up to 27.7 months
Population: Full Analysis Set (FAS) included all participants who were administered at least 1 dose of berzosertib.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Safety run-in Part (DL2) + Main Part: Berzosertib 210 mg/m^2 + Topotecan 1.25 mg/m^2
Number analyzed (Participants) | 73
months | 6.4 [4.2 to 7.6]

10. Secondary Outcome: Main Part: Change From Baseline in Physical Functioning Measured by European Organization for the Research and Treatment of Cancer Quality of Life Questionnaire (EORTC QLQ-C30)
Description: The EORTC QLQ-C30 is a participant completed 30 item questionnaire that is composed of both multi-item scales and single-item measures. These include five functional scales, three symptom scales, six single items and a global health status/QoL scale. For the physical functioning scale, subjects self-rated levels of difficulty in doing strenuous activities, taking a walk, how much they needed to stay in bed or a chair, or needed help with eating, dressing, bathing, using the toilet. The physical functioning scale had 4 possible scores (1=not at all, 2=a little, 3=quite a bit, 4=very much). Scores were averaged and transformed to 0 to 100. Higher scores indicate better functioning. A positive change from baseline indicates improvement in physical functioning.
Time Frame: Baseline (Cycle 1 Day 1), end of treatment (up to 62 weeks). Each cycle is of 21 days
Population: Full Analysis Set (FAS) included all participants who were administered at least 1 dose of berzosertib. Here, "Overall Number of Participants Analyzed" signifies those participants who were evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Safety run-in Part (DL2) + Main Part: Berzosertib 210 mg/m^2 + Topotecan 1.25 mg/m^2
Number analyzed (Participants) | 33
score on a scale | -4.0 (20.67)

11. Secondary Outcome: Main Part: Number of Participants Who Improved, Worsened or Remained Stable in European Organization for the Research and Treatment of Cancer Quality of Life and Lung Cancer Specific Questionnaire (EORTC QLQ-LC13)
Description: EORTC QLQ-LC13 is the lung cancer module of EORTC QLQ-C30 and includes questions specific to the disease associated symptoms (dyspnea, cough, hemoptysis, and site specific pain), treatment-related symptoms (sore mouth, dysphagia, neuropathy and alopecia), and analgesic use of lung cancer patients. The scale was transformed to a range of 0 to 100 using standard EORTC algorithm. Higher score indicates worse symptoms, and improvement was defined as a decrease of at least 10 points, worsening was defined as an increase of at least 10 points. All scales which had not improved nor worsened were considered stable.
Time Frame: Baseline (Cycle 1 Day 1), end of treatment (up to 62 weeks). Each cycle is of 21 days
Population: as for outcome 10
Measure: Count of Participants; unit: Participants
Arm/Group | Safety run-in Part (DL2) + Main Part: Berzosertib 210 mg/m^2 + Topotecan 1.25 mg/m^2
Number analyzed (Participants) | 33
Participants
  Improvement in Cough | 6
  Stable in Cough | 20
  Worsened in Cough | 7
  Improvement in Chest Pain | 7
  Stable in Chest Pain | 22
  Worsened in Chest Pain | 4

12. Secondary Outcome: Main Part: Change From Baseline in Health State as Measured by Visual Analogue Scale (VAS) Component of European Quality of Life 5-dimensions 5 Level Scale (EQ-5D-5L)
Description: EQ-5D-5L is comprised of the following 5 participant-reported dimensions: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. Each dimension has 5 levels: no problems, slight problems, moderate problems, severe problems, and extreme problems. The responses are used to derive overall score using a visual analog scale (VAS) that ranged from 0 to 100, where 0 is the worst health you can imagine and 100 is the best health you can imagine.
Time Frame: Baseline (Cycle 1 Day 1), end of treatment (up to 62 weeks). Each cycle is of 21 days
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Safety run-in Part (DL2) + Main Part: Berzosertib 210 mg/m^2 + Topotecan 1.25 mg/m^2
Number analyzed (Participants) | 31
score on a scale | -6.3 (19.67)

13. Secondary Outcome: Main Part: Number of Participants With Treatment-Emergent Adverse Events (TEAEs) and Treatment-Related TEAEs
Description: as for outcome 3
Time Frame: Time from first administration of study treatment up to 27.7 months
Population: Safety (SAF) Analysis Set included all participants who were administered at least 1 dose of berzosertib.
Measure: Count of Participants; unit: Participants
Arm/Group | Safety run-in Part (DL2) + Main Part: Berzosertib 210 mg/m^2 + Topotecan 1.25 mg/m^2
Number analyzed (Participants) | 73
Participants
  TEAEs | 73
  Treatment Related TEAEs | 67

14. Secondary Outcome: Main Part: Number of Participants With Clinically Significant Changes From Baseline in Vital Signs
Description: as for outcome 4
Time Frame: Time from first administration of study treatment up to 27.7 months
Population: Safety (SAF) Analysis Set included all participants who were administered at least 1 dose of berzosertib.
Measure: Count of Participants; unit: Participants
Arm/Group | Safety run-in Part (DL2) + Main Part: Berzosertib 210 mg/m^2 + Topotecan 1.25 mg/m^2
Number analyzed (Participants) | 73
Participants | 0

15. Secondary Outcome: Main Part: Number of Participants With Clinically Significant Changes From Baseline in 12-Lead Electrocardiogram (ECG) Findings
Description: as for outcome 5
Time Frame: Time from first administration of study treatment up to 27.7 months
Population: Safety (SAF) Analysis Set included all participants who were administered at least 1 dose of berzosertib.
Measure: Count of Participants; unit: Participants
Arm/Group | Safety run-in Part (DL2) + Main Part: Berzosertib 210 mg/m^2 + Topotecan 1.25 mg/m^2
Number analyzed (Participants) | 73
Participants | 0

16. Secondary Outcome: Main Part: Number of Participants With Clinically Significant Abnormalities in Laboratory Values Reported as Treatment Emergent Adverse Events (TEAEs)
Description: The laboratory measurements included hematology and biochemistry. Number of participants with clinically significant abnormalities with Grade greater than or equals to (>=) 3 in laboratory values reported as TEAEs as per NCI-CTCAE, v5.0 graded from Grade 1 to 5. Grade 1: Mild; Grade 2: Moderate; Grade 3: Severe; Grade 4: Life-threatening; Grade 5: Death. Clinically Significance was decided by investigator. The laboratory assessments were graded according to NCI-CTCAE version 5.0 and data for individual clinically significant abnormalities (Grade >= 3) was extracted using data source (ADLBHEMA). The data categorized here may not necessarily be considered as TEAE by the investigator during the reporting of TEAEs and there is no correlation between the grade >=3 treatment related TEAEs hematology parameters and the TEAEs in the AE module.
Time Frame: Time from first administration of study treatment up to 27.7 months
Population: Safety (SAF) Analysis Set included all participants who were administered at least 1 dose of berzosertib.
Measure: Count of Participants; unit: Participants
Arm/Group | Safety run-in Part (DL2) + Main Part: Berzosertib 210 mg/m^2 + Topotecan 1.25 mg/m^2
Number analyzed (Participants) | 73
Participants
  Anemia | 18
  Lymphocyte count decreased | 17
  Neutrophil count decreased | 28
  Platelet count decreased | 26
  White blood cell decreased | 19
  Alanine aminotransferase increased | 2
  Alkaline phosphatase increased | 1
  Aspartate transaminase increased | 1
  Blood bilirnbin increased | 3
  Hypokalemia | 8
  Hyponatremia | 4

17. Secondary Outcome: Safety Run-in Part: Objective Response Rate According to Response Evaluation Criteria in Solid Tumors (RECIST) Version 1.1 as Assessed by Investigator
Description: as for outcome 1
Time Frame: Time from first administration of study treatment up to 27.7 months
Population: Full Analysis Set (FAS) included all participants who were administered at least 1 dose of berzosertib.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Safety run-in Part (DL 1): Berzosertib 105 mg/m^2 + Topotecan 1.25 mg/m^2 | Safety run-in Part (DL2) + Main Part: Berzosertib 210 mg/m^2 + Topotecan 1.25 mg/m^2
Number analyzed (Participants) | 3 | 3
percentage of participants | 33.3 [0.8 to 90.6] | 0.0 [0.0 to 70.8]

18. Secondary Outcome: Safety Run-in Part: Duration of Response (DoR) According to Response Evaluation Criteria in Solid Tumors (RECIST) Version 1.1 as Assessed by Investigator
Description: as for outcome 7
Time Frame: Time from first administration of study treatment up to 27.7 months
Population: as for outcome 10
Measure: Number; unit: months
Arm/Group | Safety run-in Part (DL 1): Berzosertib 105 mg/m^2 + Topotecan 1.25 mg/m^2 | Safety run-in Part (DL2) + Main Part: Berzosertib 210 mg/m^2 + Topotecan 1.25 mg/m^2
Number analyzed (Participants) | 1 | 0
months | 7.2 |

19. Secondary Outcome: Safety Run-in Part: Progression-free Survival (PFS) According to Response Evaluation Criteria in Solid Tumors (RECIST) Version 1.1 as Assessed by Investigator
Description: as for outcome 8
Time Frame: as for outcome 8
Population: Full Analysis Set (FAS) included all participants who were administered at least 1 dose of berzosertib.
Measure: Median (Full Range); unit: months
Arm/Group | Safety run-in Part (DL 1): Berzosertib 105 mg/m^2 + Topotecan 1.25 mg/m^2 | Safety run-in Part (DL2) + Main Part: Berzosertib 210 mg/m^2 + Topotecan 1.25 mg/m^2
Number analyzed (Participants) | 3 | 3
months | 14.3 [4.0 to 14.3] | 3.3 [1.2 to 8.1]

20. Secondary Outcome: Safety Run-in Part: Overall Survival (OS)
Description: Overall survival is defined as the time from first administration of study treatment to the date of death.
Time Frame: Time from first administration of study treatment to the date of death, assessed up to 27.7 months
Population: Full Analysis Set (FAS) included all participants who were administered at least 1 dose of berzosertib.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Safety run-in Part (DL 1): Berzosertib 105 mg/m^2 + Topotecan 1.25 mg/m^2 | Safety run-in Part (DL2) + Main Part: Berzosertib 210 mg/m^2 + Topotecan 1.25 mg/m^2
Number analyzed (Participants) | 3 | 3
months | NA [8.0 to NA] — Due to small number of events, median and upper limit of 95% Confidence Interval from Kaplan-Meier survival curves could not be derived. | 15.3 [10.0 to NA] — Due to small number of events, upper limit of 95% Confidence Interval from Kaplan-Meier survival curves could not be derived.

21. Secondary Outcome: Safety Run-in Part: Change From Baseline in Physical Functioning Measured by European Organization for the Research and Treatment of Cancer Quality of Life Questionnaire (EORTC QLQ-C30)
Description: as for outcome 10
Time Frame: Baseline (Cycle 1 Day 1), end of treatment (up to 64 weeks). Each cycle is of 21 days
Population: As per changes in planned analysis, the outcome measure related to quality of life for safety run-in part was not assessed.
Arm/Group | Safety run-in Part (DL 1): Berzosertib 105 mg/m^2 + Topotecan 1.25 mg/m^2 | Safety run-in Part (DL2) + Main Part: Berzosertib 210 mg/m^2 + Topotecan 1.25 mg/m^2
Number analyzed (Participants) | 0 | 0

22. Secondary Outcome: Safety Run-in Part: Change From Baseline in Cough, Dyspnea and Chest Pain Measured by European Organization for the Research and Treatment of Cancer Quality of Life and Lung Cancer Specific Questionnaire (EORTC QLQ-LC13)
Description: EORTC QLQ-LC13 consisted of 13 questions relating to disease symptoms specific to lung cancer and treatment side effects typical of treatment with chemotherapy and radiotherapy. The EORTC QLQ-LC13 module generated one multiple-item score assessing dyspnea and a series of single item scores assessing coughing, hemoptysis, sore mouth, dysphagia, peripheral neuropathy, alopecia, pain in chest, pain in arms or shoulder and pain in other parts. Score range: 0 (no burden of symptom domain or single symptom item) to 100 (highest burden of symptoms for symptom domains and single items).
Time Frame: Baseline (Cycle 1 Day 1), end of treatment (up to 64 weeks). Each cycle is of 21 days
Population: as for outcome 21
Arm/Group | Safety run-in Part (DL 1): Berzosertib 105 mg/m^2 + Topotecan 1.25 mg/m^2 | Safety run-in Part (DL2) + Main Part: Berzosertib 210 mg/m^2 + Topotecan 1.25 mg/m^2
Number analyzed (Participants) | 0 | 0

23. Secondary Outcome: Safety Run-in Part: Change From Baseline in Health State as Measured by Visual Analogue Scale (VAS) Component of European Quality of Life 5-dimensions 5 Level Scale (EQ-5D-5L)
Description: as for outcome 12
Time Frame: Baseline (Cycle 1 Day 1), end of treatment (up to 64 weeks). Each cycle is of 21 days
Population: as for outcome 21
Groups:
- Safety run-in Part (DL 1): Berzosertib 105 mg/m^2 + Topotecan 1.25 mg/m^2: Participants received Berzosertib at a dose of 105 milligrams per square meter (mg/m^2 ) intravenously on Day 2 and Day 5 of each 21-day cycle in combination with Topotecan at a dose of 1.25 mg/m^2 intravenously on Days 1 through 5 of each 21-day cycle in DL1 of safety run-in part until disease progression or other criteria for study intervention discontinuation are met.
Arm/Group | Safety run-in Part (DL 1): Berzosertib 105 mg/m^2 + Topotecan 1.25 mg/m^2 | Safety run-in Part (DL2) + Main Part: Berzosertib 210 mg/m^2 + Topotecan 1.25 mg/m^2
Number analyzed (Participants) | 0 | 0

24. Secondary Outcome: Safety Run-in Part: Area Under the Plasma Concentration-Time Curve From Time Zero to the Last Sampling Time (AUC0-tlast) of Berzosertib
Description: Area under the plasma concentration versus time curve from time zero to the last sampling time t at which the concentration was at or above the lower limit of quantification (LLOQ). AUC0-t was calculated according to the mixed log-linear trapezoidal rule.
Time Frame: Pre-dose, 1, 2, 3, 4, 8, 24, 48 and 72 hours after dose on Cycle 1 Day 2 (each cycle is of 21 days)
Population: Pharmacokinetic Analysis Set (PKS) included all participants who were administered at least 1 complete infusion of berzosertib in the Safety Run-in Part in Japan and for whom at least 1 quantifiable post-dose plasma concentration of berzosertib was obtained.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hour*nanogram per milliliter (h*ng/mL)
Arm/Group | Safety run-in Part (DL 1): Berzosertib 105 mg/m^2 + Topotecan 1.25 mg/m^2 | Safety run-in Part (DL2) + Main Part: Berzosertib 210 mg/m^2 + Topotecan 1.25 mg/m^2
Number analyzed (Participants) | 3 | 3
hour*nanogram per milliliter (h*ng/mL) | 2330 (0.8) | 4090 (7.1)

25. Secondary Outcome: Safety Run-in Part: Dose Normalized Area Under the Plasma Concentration-Time Curve From Time Zero to the Last Sampling Time (AUC0-tlast/Dose) of Berzosertib
Description: AUC0-t/Dose was defined as AUC from time of dosing to the time of the last measurable concentration divided by dose. AUC0-t/dose was measured in hour*nanogram per milliliter per milligram (h*ng/mL/mg).
Time Frame: Pre-dose, 1, 2, 3, 4, 8, 24, 48 and 72 hours after dose on Cycle 1 Day 2 (each cycle is of 21 days)
Population: as for outcome 24
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL/mg
Arm/Group | Safety run-in Part (DL 1): Berzosertib 105 mg/m^2 + Topotecan 1.25 mg/m^2 | Safety run-in Part (DL2) + Main Part: Berzosertib 210 mg/m^2 + Topotecan 1.25 mg/m^2
Number analyzed (Participants) | 3 | 3
h*ng/mL/mg | 12.2 (9.9) | 11.1 (9.8)

26. Secondary Outcome: Safety Run-in Part: Area Under the Plasma Concentration-Time Curve From Time Zero Extrapolated to Infinity (AUC0-inf) of Berzosertib
Description: AUC0-inf was calculated by combining AUC0-t and AUCextra. AUCextra represents an extrapolated value obtained by Clast pred/Lambda z, where Clast pred was the calculated plasma concentration at the last sampling time point at which the measured plasma concentration is at or above the Lower Limit of quantification (LLOQ) and Lambda z was the apparent terminal rate constant determined by log-linear regression analysis of the measured plasma concentrations of the terminal log-linear phase.
Time Frame: Pre-dose, 1, 2, 3, 4, 8, 24, 48 and 72 hours after dose on Cycle 1 Day 2 (each cycle is of 21 days)
Population: as for outcome 24
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | Safety run-in Part (DL 1): Berzosertib 105 mg/m^2 + Topotecan 1.25 mg/m^2 | Safety run-in Part (DL2) + Main Part: Berzosertib 210 mg/m^2 + Topotecan 1.25 mg/m^2
Number analyzed (Participants) | 3 | 3
h*ng/mL | 2460 (1.4) | 4310 (8.8)

27. Secondary Outcome: Safety Run-in Part: Dose Normalized Area Under the Plasma Concentration-Time Curve From Time Zero Extrapolated to Infinity (AUC0-inf/Dose) of Berzosertib
Description: AUC0-inf/Dose was defined as AUC extrapolated to infinity divided by dose.
Time Frame: Pre-dose, 1, 2, 3, 4, 8, 24, 48 and 72 hours after dose on Cycle 1 Day 2 (each cycle is of 21 days)
Population: as for outcome 24
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL/mg
Arm/Group | Safety run-in Part (DL 1): Berzosertib 105 mg/m^2 + Topotecan 1.25 mg/m^2 | Safety run-in Part (DL2) + Main Part: Berzosertib 210 mg/m^2 + Topotecan 1.25 mg/m^2
Number analyzed (Participants) | 3 | 3
h*ng/mL/mg | 12.8 (11.0) | 11.7 (11.4)

28. Secondary Outcome: Safety Run-in Part: Area Under the Plasma Concentration-Time Curve From Time Zero to 48 Hours (AUC0-48h) of Berzosertib
Description: Area under the concentration-time curve from pre-dose (time 0) to 48 hours post-dose calculated using the linear-log trapezoidal rule
Time Frame: Pre-dose, 1, 2, 3, 4, 8, 24 and 48 hours after dose on Cycle 1 Day 2 (each cycle is of 21 days)
Population: as for outcome 24
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | Safety run-in Part (DL 1): Berzosertib 105 mg/m^2 + Topotecan 1.25 mg/m^2 | Safety run-in Part (DL2) + Main Part: Berzosertib 210 mg/m^2 + Topotecan 1.25 mg/m^2
Number analyzed (Participants) | 3 | 3
h*ng/mL | 2160 (2.0) | 3790 (5.6)

29. Secondary Outcome: Safety Run-in Part: Dose Normalized Area Under the Plasma Concentration-Time Curve From Time Zero to 48 Hours (AUC0-48h/Dose) of Berzosertib
Description: AUC0-48 hour/Dose was defined as AUC from time of dosing to 48 hours divided by dose.
Time Frame: Pre-dose, 1, 2, 3, 4, 8, 24 and 48 hours after dose on Cycle 1 Day 2 (each cycle is of 21 days)
Population: as for outcome 24
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL/mg
Arm/Group | Safety run-in Part (DL 1): Berzosertib 105 mg/m^2 + Topotecan 1.25 mg/m^2 | Safety run-in Part (DL2) + Main Part: Berzosertib 210 mg/m^2 + Topotecan 1.25 mg/m^2
Number analyzed (Participants) | 3 | 3
h*ng/mL/mg | 11.3 (9.7) | 10.3 (8.7)

30. Secondary Outcome: Safety Run-in Part: Area Under the Plasma Concentration-Time Curve From Time Zero to 72 Hours (AUC0-72h) of Berzosertib
Description: Area under the concentration-time curve from pre-dose (time 0) to 72 hours post-dose calculated using the linear-log trapezoidal rule
Time Frame: Pre-dose, 1, 2, 3, 4, 8, 24, 48 and 72 hours after dose on Cycle 1 Day 2 (each cycle is of 21 days)
Population: as for outcome 24
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | Safety run-in Part (DL 1): Berzosertib 105 mg/m^2 + Topotecan 1.25 mg/m^2 | Safety run-in Part (DL2) + Main Part: Berzosertib 210 mg/m^2 + Topotecan 1.25 mg/m^2
Number analyzed (Participants) | 3 | 3
h*ng/mL | 2340 (0.8) | 4110 (7.1)

31. Secondary Outcome: Safety Run-in Part: Dose Normalized Area Under the Plasma Concentration-Time Curve From Time Zero to 72 Hours (AUC0-72h/Dose) of Berzosertib
Description: AUC0-72 hour/Dose was defined as AUC from time of dosing to 72 hours divided by dose.
Time Frame: Pre-dose, 1, 2, 3, 4, 8, 24, 48 and 72 hours after dose on Cycle 1 Day 2 (each cycle is of 21 days)
Population: as for outcome 24
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL/mg
Arm/Group | Safety run-in Part (DL 1): Berzosertib 105 mg/m^2 + Topotecan 1.25 mg/m^2 | Safety run-in Part (DL2) + Main Part: Berzosertib 210 mg/m^2 + Topotecan 1.25 mg/m^2
Number analyzed (Participants) | 3 | 3
h*ng/mL/mg | 12.2 (9.9) | 11.2 (9.9)

32. Secondary Outcome: Safety Run-in Part: Maximum Observed Plasma Concentration (Cmax) of Berzosertib
Description: Cmax was obtained directly from the plasma concentration versus time curve.
Time Frame: Pre-dose, 1, 2, 3, 4, 8, 24, 48 and 72 hours after dose on Cycle 1 Day 2 (each cycle is of 21 days)
Population: as for outcome 24
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Safety run-in Part (DL 1): Berzosertib 105 mg/m^2 + Topotecan 1.25 mg/m^2 | Safety run-in Part (DL2) + Main Part: Berzosertib 210 mg/m^2 + Topotecan 1.25 mg/m^2
Number analyzed (Participants) | 3 | 3
ng/mL | 259 (23.5) | 446 (17.7)

33. Secondary Outcome: Safety Run-in Part: Dose Normalized Maximum Observed Plasma Concentration (Cmax/Dose) of Berzosertib
Description: Dose normalized was calculated as Cmax obtained directly from the concentration versus time curve divided by dose. Cmax/dose was measured in nanogram per milliliter per milligram (ng/mL/mg).
Time Frame: Pre-dose, 1, 2, 3, 4, 8, 24, 48 and 72 hours after dose on Cycle 1 Day 2 (each cycle is of 21 days)
Population: as for outcome 24
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL/mg
Arm/Group | Safety run-in Part (DL 1): Berzosertib 105 mg/m^2 + Topotecan 1.25 mg/m^2 | Safety run-in Part (DL2) + Main Part: Berzosertib 210 mg/m^2 + Topotecan 1.25 mg/m^2
Number analyzed (Participants) | 3 | 3
ng/mL/mg | 1.35 (27.5) | 1.21 (24.9)

34. Secondary Outcome: Safety Run-in Part: Plasma Observed Concentration at the End of the Infusion (Ceoi) of Berzosertib
Description: Ceoi was the observed concentration at the end of the infusion period. This was taken directly from the observed Berzosetib concentration-time data.
Time Frame: Pre-dose, 1, 2, 3, 4, 8, 24, 48 and 72 hours after dose on Cycle 1 Day 2; Pre-dose, 1 and 1.5 hours after dose on Cycle 1 Day 5 (each cycle is of 21 days)
Population: as for outcome 24
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Safety run-in Part (DL 1): Berzosertib 105 mg/m^2 + Topotecan 1.25 mg/m^2 | Safety run-in Part (DL2) + Main Part: Berzosertib 210 mg/m^2 + Topotecan 1.25 mg/m^2
Number analyzed (Participants) | 3 | 3
ng/mL
  Cycle 1 Day 2 | 259 (23.5) | 446 (17.7)
  Cycle 1 Day 5 | 341 (23.1) | 500 (42.7)

35. Secondary Outcome: Safety Run-in Part: Plasma Observed Concentration Immediately Before Next Dosing (Ctrough) of Berzosertib
Description: Ctrough was the plasma concentration observed immediately before next dosing.
Time Frame: Pre-dose on Cycle 1 Day 5 (each cycle is of 21 days)
Population: as for outcome 24
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Safety run-in Part (DL 1): Berzosertib 105 mg/m^2 + Topotecan 1.25 mg/m^2 | Safety run-in Part (DL2) + Main Part: Berzosertib 210 mg/m^2 + Topotecan 1.25 mg/m^2
Number analyzed (Participants) | 3 | 3
ng/mL | 4.84 (22.3) | 8.57 (23.6)

36. Secondary Outcome: Safety Run-in Part: Apparent Total Body Clearance (CL) of Berzosertib
Description: CL was a measure of the rate at which a drug was metabolized or eliminated by normal biological processes. CL was calculated as Dose/AUC0-inf, where AUC0-inf was estimated by determining the total area under the curve of the concentration versus time curve extrapolated to infinity. AUC0-inf was calculated as AUC0-t + Clast pred/Lambda Z, where Clast pred was the calculated plasma concentration at the last sampling time point at which the measured plasma concentration was at or above the lower limit of quantification (LLQ) and Lambda Z was the apparent terminal rate constant determined from the terminal slope of the log-transformed plasma concentration curve.
Time Frame: Pre-dose, 1, 2, 3, 4, 8, 24, 48 and 72 hours after dose on Cycle 1 Day 2 (each cycle is of 21 days)
Population: as for outcome 24
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: liter per hour
Arm/Group | Safety run-in Part (DL 1): Berzosertib 105 mg/m^2 + Topotecan 1.25 mg/m^2 | Safety run-in Part (DL2) + Main Part: Berzosertib 210 mg/m^2 + Topotecan 1.25 mg/m^2
Number analyzed (Participants) | 3 | 3
liter per hour | 77.8 (11.0) | 85.4 (11.4)

37. Secondary Outcome: Safety Run-in Part: Accumulation Ratio for Maximum Observed Plasma Concentration [Racc(Cmax)] of Berzosertib
Description: Accumulation ratio of Cmax was calculated as Cmax after dosing on Day 5 divided by Cmax after dosing on Day 2 of Cycle 1.
Time Frame: as for outcome 34
Population: as for outcome 24
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ratio
Arm/Group | Safety run-in Part (DL 1): Berzosertib 105 mg/m^2 + Topotecan 1.25 mg/m^2 | Safety run-in Part (DL2) + Main Part: Berzosertib 210 mg/m^2 + Topotecan 1.25 mg/m^2
Number analyzed (Participants) | 3 | 3
ratio | 1.32 (16.3) | 1.12 (24.9)

38. Secondary Outcome: Safety Run-in Part: Time to Reach the Maximum Observed Plasma Concentration (Tmax) of Berzosertib
Description: Tmax was obtained directly from the plasma concentration versus time curve.
Time Frame: Pre-dose, 1, 2, 3, 4, 8, 24, 48 and 72 hours after dose on Cycle 1 Day 2 (each cycle is of 21 days)
Population: as for outcome 24
Measure: Median (Full Range); unit: hours
Arm/Group | Safety run-in Part (DL 1): Berzosertib 105 mg/m^2 + Topotecan 1.25 mg/m^2 | Safety run-in Part (DL2) + Main Part: Berzosertib 210 mg/m^2 + Topotecan 1.25 mg/m^2
Number analyzed (Participants) | 3 | 3
hours | 1.17 [1.13 to 1.2] | 1.20 [1.17 to 1.23]

39. Secondary Outcome: Safety Run-in Part: Apparent Terminal Half-life (t1/2) of Berzosertib
Description: T1/2 was defined as the time required for the concentration or amount of drug in the body to be reduced by one-half. T1/2 was calculated by natural log 2 divided by Lambda z. Lambda z was determined from the terminal slope of the log-transformed plasma concentration curve using linear regression method.
Time Frame: Pre-dose, 1, 2, 3, 4, 8, 24, 48 and 72 hours after dose on Cycle 1 Day 2 (each cycle is of 21 days)
Population: as for outcome 24
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hours
Arm/Group | Safety run-in Part (DL 1): Berzosertib 105 mg/m^2 + Topotecan 1.25 mg/m^2 | Safety run-in Part (DL2) + Main Part: Berzosertib 210 mg/m^2 + Topotecan 1.25 mg/m^2
Number analyzed (Participants) | 3 | 3
hours | 17.6 (10.1) | 17.0 (13.5)

40. Secondary Outcome: Safety Run-in Part: Last Sampling Time (Tlast) of Berzosertib
Description: tlast is defined as the last sampling time at which the concentration is at or above the lower limit of quantification.
Time Frame: Pre-dose, 1, 2, 3, 4, 8, 24, 48 and 72 hours after dose on Cycle 1 Day 2 (each cycle is of 21 days)
Population: as for outcome 24
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hours
Arm/Group | Safety run-in Part (DL 1): Berzosertib 105 mg/m^2 + Topotecan 1.25 mg/m^2 | Safety run-in Part (DL2) + Main Part: Berzosertib 210 mg/m^2 + Topotecan 1.25 mg/m^2
Number analyzed (Participants) | 3 | 3
hours | 70.4 (0.3) | 70.6 (0.7)

41. Secondary Outcome: Safety Run-in Part: Apparent Volume of Distribution During Terminal Phase (Vz) of Berzosertib
Description: Vz: the distribution of a study drug between plasma and the rest of the body after oral dosing. For single dose Vz = Dose/(AUC0-inf*Lambda Z), where AUC0-inf = (AUC0-t + Clast pred/Lambda Z). Clastpred was the calculated plasma concentration at the last sampling time point at which the measured plasma concentration was at or above the LLOQ and Lambda Z = the apparent terminal rate constant determined from the terminal slope of the log-transformed plasma concentration curve.
Time Frame: Pre-dose, 1, 2, 3, 4, 8, 24, 48 and 72 hours after dose on Cycle 1 Day 2 (each cycle is of 21 days)
Population: as for outcome 24
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: liters
Arm/Group | Safety run-in Part (DL 1): Berzosertib 105 mg/m^2 + Topotecan 1.25 mg/m^2 | Safety run-in Part (DL2) + Main Part: Berzosertib 210 mg/m^2 + Topotecan 1.25 mg/m^2
Number analyzed (Participants) | 3 | 3
liters | 1980 (4.2) | 2100 (5.8)

ADVERSE EVENTS:
Time Frame: Time from first administration of study treatment up to 27.7 months
Arm/Group | Safety run-in Part (Dose Level 1 [DL 1]): Berzosertib 105 mg/m^2 + Topotecan 1.25 mg/m^2 | Safety run-in Part (DL2) + Main Part: Berzosertib 210 mg/m^2 + Topotecan 1.25 mg/m^2
All-Cause Mortality (participants affected / at risk) | 1/3 | 63/73
Serious Adverse Events (participants affected / at risk) | 0/3 | 31/73
Other Adverse Events (participants affected / at risk) | 3/3 | 70/73
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Safety run-in Part (Dose Level 1 [DL 1]): Berzosertib 105 mg/m^2 + Topotecan 1.25 mg/m^2 (N=3) | Safety run-in Part (DL2) + Main Part: Berzosertib 210 mg/m^2 + Topotecan 1.25 mg/m^2 (N=73)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 4 (5)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 4 (4)
Myelosuppression (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 3 (4)
Acute coronary syndrome (Cardiac disorders) | 0 (0) | 1 (1)
Vestibular disorder (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 2 (2)
Asthenia (General disorders) | 0 (0) | 1 (1)
Disease progression (General disorders) | 0 (0) | 1 (1)
Fatigue (General disorders) | 0 (0) | 1 (1)
General physical health deterioration (General disorders) | 0 (0) | 1 (1)
Multiple organ dysfunction syndrome (General disorders) | 0 (0) | 1 (2)
Pyrexia (General disorders) | 0 (0) | 1 (1)
Liver injury (Hepatobiliary disorders) | 0 (0) | 2 (3)
COVID-19 (Infections and infestations) | 0 (0) | 4 (4)
COVID-19 pneumonia (Infections and infestations) | 0 (0) | 3 (3)
Enterococcal sepsis (Infections and infestations) | 0 (0) | 1 (1)
Lung abscess (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia bacterial (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia pneumococcal (Infections and infestations) | 0 (0) | 1 (1)
Sepsis (Infections and infestations) | 0 (0) | 2 (2)
Septic shock (Infections and infestations) | 0 (0) | 1 (1)
Serratia sepsis (Infections and infestations) | 0 (0) | 1 (1)
Staphylococcal sepsis (Infections and infestations) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (3)
Urosepsis (Infections and infestations) | 0 (0) | 1 (1)
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Neutrophil count decreased (Investigations) | 0 (0) | 2 (2)
Platelet count decreased (Investigations) | 0 (0) | 2 (3)
White blood cell count decreased (Investigations) | 0 (0) | 1 (1)
Hypoglycaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 0 (0) | 1 (1)
Seizure (Nervous system disorders) | 0 (0) | 1 (1)
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 6 (7)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Safety run-in Part (Dose Level 1 [DL 1]): Berzosertib 105 mg/m^2 + Topotecan 1.25 mg/m^2 (N=3) | Safety run-in Part (DL2) + Main Part: Berzosertib 210 mg/m^2 + Topotecan 1.25 mg/m^2 (N=73)
Anaemia (Blood and lymphatic system disorders) | 3 (6) | 48 (89)
Coagulopathy (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Leukopenia (Blood and lymphatic system disorders) | 1 (1) | 2 (2)
Myelosuppression (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Neutropenia (Blood and lymphatic system disorders) | 1 (1) | 23 (37)
Thrombocytopenia (Blood and lymphatic system disorders) | 3 (3) | 26 (45)
Thrombocytosis (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Arrhythmia (Cardiac disorders) | 0 (0) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 2 (2)
Cardiac failure (Cardiac disorders) | 0 (0) | 1 (1)
Sinus tachycardia (Cardiac disorders) | 0 (0) | 1 (1)
Tachycardia (Cardiac disorders) | 0 (0) | 3 (5)
Vestibular disorder (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Hypothyroidism (Endocrine disorders) | 0 (0) | 1 (1)
Immune-mediated hypothyroidism (Endocrine disorders) | 0 (0) | 1 (1)
Conjunctival pallor (Eye disorders) | 0 (0) | 1 (1)
Diplopia (Eye disorders) | 0 (0) | 1 (1)
Eye discharge (Eye disorders) | 0 (0) | 1 (1)
Macular oedema (Eye disorders) | 0 (0) | 1 (1)
Abdominal discomfort (Gastrointestinal disorders) | 0 (0) | 1 (2)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 3 (3)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 2 (2)
Constipation (Gastrointestinal disorders) | 1 (1) | 13 (16)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 11 (12)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Flatulence (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 3 (5)
Gingival pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
Haemorrhoids (Gastrointestinal disorders) | 0 (0) | 1 (1)
Haemorrhoids thrombosed (Gastrointestinal disorders) | 0 (0) | 1 (1)
Lip dry (Gastrointestinal disorders) | 0 (0) | 1 (1)
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (2) | 20 (29)
Oral disorder (Gastrointestinal disorders) | 0 (0) | 1 (1)
Tooth loss (Gastrointestinal disorders) | 0 (0) | 1 (1)
Toothache (Gastrointestinal disorders) | 1 (2) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 10 (11)
Asthenia (General disorders) | 0 (0) | 18 (31)
Chest discomfort (General disorders) | 0 (0) | 2 (2)
Chest pain (General disorders) | 0 (0) | 1 (2)
Chills (General disorders) | 0 (0) | 2 (2)
Face oedema (General disorders) | 0 (0) | 1 (1)
Fatigue (General disorders) | 1 (1) | 10 (12)
Gait disturbance (General disorders) | 0 (0) | 1 (1)
Generalised oedema (General disorders) | 0 (0) | 1 (2)
Hyperthermia (General disorders) | 0 (0) | 1 (1)
Influenza like illness (General disorders) | 0 (0) | 1 (1)
Injection site pruritus (General disorders) | 0 (0) | 1 (1)
Localised oedema (General disorders) | 0 (0) | 2 (2)
Malaise (General disorders) | 0 (0) | 4 (4)
Mucosal inflammation (General disorders) | 0 (0) | 4 (4)
Oedema peripheral (General disorders) | 0 (0) | 3 (3)
Pain (General disorders) | 0 (0) | 2 (2)
Pyrexia (General disorders) | 0 (0) | 5 (9)
Secretion discharge (General disorders) | 0 (0) | 1 (1)
Swelling face (General disorders) | 0 (0) | 1 (1)
Cholestasis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Hepatic pain (Hepatobiliary disorders) | 0 (0) | 1 (1)
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 (0) | 1 (1)
Liver injury (Hepatobiliary disorders) | 0 (0) | 3 (3)
Hypersensitivity (Immune system disorders) | 0 (0) | 1 (1)
Bronchiolitis (Infections and infestations) | 0 (0) | 1 (1)
Bronchitis (Infections and infestations) | 0 (0) | 1 (1)
COVID-19 (Infections and infestations) | 1 (1) | 4 (4)
Candida infection (Infections and infestations) | 0 (0) | 1 (1)
Diverticulitis (Infections and infestations) | 0 (0) | 1 (1)
Gastroenteritis (Infections and infestations) | 0 (0) | 1 (5)
Herpes zoster reactivation (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 0 (0) | 8 (9)
Respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1)
Sinusitis (Infections and infestations) | 0 (0) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 2 (3)
Wound infection (Infections and infestations) | 0 (0) | 1 (1)
Compression fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Infusion related reaction (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Radiation oesophagitis (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Radiation pneumonitis (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Spinal fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Activated partial thromboplastin time prolonged (Investigations) | 0 (0) | 2 (4)
Alanine aminotransferase increased (Investigations) | 0 (0) | 7 (7)
Amylase increased (Investigations) | 0 (0) | 2 (4)
Aspartate aminotransferase decreased (Investigations) | 0 (0) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 7 (7)
Blood albumin decreased (Investigations) | 0 (0) | 2 (2)
Blood alkaline phosphatase increased (Investigations) | 0 (0) | 6 (8)
Blood bilirubin increased (Investigations) | 0 (0) | 2 (2)
Blood cholesterol increased (Investigations) | 0 (0) | 1 (1)
Blood creatinine increased (Investigations) | 0 (0) | 3 (4)
Blood glucose increased (Investigations) | 0 (0) | 1 (2)
Blood lactate dehydrogenase increased (Investigations) | 0 (0) | 2 (2)
Blood lactic acid increased (Investigations) | 0 (0) | 1 (1)
Blood magnesium decreased (Investigations) | 0 (0) | 2 (2)
Blood phosphorus decreased (Investigations) | 0 (0) | 1 (2)
Blood sodium decreased (Investigations) | 0 (0) | 1 (1)
Blood urea increased (Investigations) | 0 (0) | 1 (1)
C-reactive protein increased (Investigations) | 0 (0) | 1 (1)
CD4/CD8 ratio decreased (Investigations) | 0 (0) | 1 (1)
Creatinine renal clearance decreased (Investigations) | 0 (0) | 1 (1)
Electrocardiogram QT prolonged (Investigations) | 1 (1) | 1 (1)
Gamma-glutamyltransferase increased (Investigations) | 0 (0) | 4 (5)
Haemoglobin decreased (Investigations) | 0 (0) | 2 (2)
Lipase increased (Investigations) | 1 (1) | 6 (8)
Lymphocyte count decreased (Investigations) | 0 (0) | 9 (21)
Neutrophil count decreased (Investigations) | 0 (0) | 12 (18)
Platelet count decreased (Investigations) | 0 (0) | 22 (45)
Platelet count increased (Investigations) | 0 (0) | 1 (1)
Urine output decreased (Investigations) | 0 (0) | 1 (1)
Weight decreased (Investigations) | 0 (0) | 6 (8)
White blood cell count decreased (Investigations) | 0 (0) | 13 (22)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 18 (22)
Electrolyte imbalance (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Gout (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 4 (4)
Hyperkalaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 (0) | 7 (8)
Hypocalcaemia (Metabolism and nutrition disorders) | 0 (0) | 6 (8)
Hypochloraemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 8 (9)
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 (0) | 4 (5)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 5 (11)
Hypophosphataemia (Metabolism and nutrition disorders) | 0 (0) | 3 (4)
Malnutrition (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Disturbance in attention (Nervous system disorders) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 0 (0) | 5 (6)
Dysgeusia (Nervous system disorders) | 1 (1) | 3 (3)
Headache (Nervous system disorders) | 0 (0) | 7 (8)
Hemianopia homonymous (Nervous system disorders) | 0 (0) | 1 (1)
Hemiparesis (Nervous system disorders) | 0 (0) | 1 (1)
Memory impairment (Nervous system disorders) | 0 (0) | 1 (1)
Neuropathy peripheral (Nervous system disorders) | 1 (1) | 2 (2)
Paraesthesia (Nervous system disorders) | 0 (0) | 2 (2)
Presyncope (Nervous system disorders) | 0 (0) | 1 (1)
Seizure (Nervous system disorders) | 0 (0) | 1 (1)
Transient aphasia (Nervous system disorders) | 0 (0) | 1 (1)
Tremor (Nervous system disorders) | 0 (0) | 1 (1)
Device malfunction (Product Issues) | 0 (0) | 1 (1)
Anxiety (Psychiatric disorders) | 0 (0) | 2 (2)
Confusional state (Psychiatric disorders) | 0 (0) | 1 (1)
Depression (Psychiatric disorders) | 0 (0) | 1 (1)
Insomnia (Psychiatric disorders) | 0 (0) | 5 (5)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 1 (1)
Choluria (Renal and urinary disorders) | 0 (0) | 1 (1)
Nephrolithiasis (Renal and urinary disorders) | 0 (0) | 1 (1)
Renal impairment (Renal and urinary disorders) | 0 (0) | 1 (1)
Aphonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 7 (8)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 11 (14)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (3)
Dyspnoea paroxysmal nocturnal (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 6 (6)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 4 (4)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Sputum discoloured (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Alopecia (Skin and subcutaneous tissue disorders) | 2 (2) | 3 (3)
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Nail disorder (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Night sweats (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)
Petechiae (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Photosensitivity reaction (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (3)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Rash pruritic (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Skin lesion (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 0 (0) | 4 (4)
Hypotension (Vascular disorders) | 0 (0) | 2 (3)
Orthostatic hypotension (Vascular disorders) | 0 (0) | 1 (1)
Pallor (Vascular disorders) | 0 (0) | 2 (2)
Phlebitis (Vascular disorders) | 0 (0) | 1 (6)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2021-06-21): https://cdn.clinicaltrials.gov/large-docs/96/NCT04768296/Prot_000.pdf
  • Statistical Analysis Plan (2023-04-17): https://cdn.clinicaltrials.gov/large-docs/96/NCT04768296/SAP_001.pdf